CLINICAL TRIAL: NCT04045223
Title: Circulating Cell-free Mitochondrial DNA Triggering Epidural Related Maternal Fever (ERMF) in Obstetric Anesthesia: a Pilot Study
Brief Title: Mitochondrial DNA Triggering Epidural Related Maternal Fever
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Ass.-Prof. PD Dr. Klaus Ulrich Klein, Principle Investigator, Klaus Ulrich Klein; MD, Medical University of Vienna
Other Study IDs: 2119/2017
Record Dates: First submitted 2019-07-25; First posted 2019-08-05 (Actual); Last update posted 2022-01-03 (Actual); Status verified 2021-12

CONDITIONS: Mitochondrial DNA; Epidural Related Maternal Fever (ERMF)
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cell-free mitochondrial DNA
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Epidural analgesia and fever: Group 1 will be patients with vaginal delivery and having an epidural analgesia that develop fever during delivery.
  Interventions: Other: Blood samples
- Epidural analgesia and no fever: Group 2 will be patients with vaginal delivery and having an epidural analgesia that do not develop fever during delivery.
  Interventions: Other: Blood samples
- No epidural analgesia: Group 3 serves as additional control group and consists of patients having no epidural analgesia and no fever.
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — Maternal blood will be taken at arrival at the delivery unit and after delivery. Furthermore, placental blood will be taken after delivery.

SUMMARY:
Background: Giving birth is a critical moment for the mother and the fetus, potentially accompanied by stress, tissue damage, cell injury, placental hypoxia and sometimes multisystem vascular syndrome known as preeclampsia. Epidural analgesia with a local anesthetic is a common anesthetic approach during labor. Local anesthetics inhibit the oxidative phosphorylation and impair the synthesis of ATP, resulting in mitochondrial dysfunction and increased reactive oxygen species. Especially when the high demand of ATP during pregnancy cannot be reached, apoptosis will occur in an anaerobic environment. During apoptosis the cell membrane integrity is disturbed, releasing the cytoplasm into the blood circulation. Circulating cell-free mitochondrial DNA acts as a damage associated molecular pattern (DAMP) by activating the innate immune system leading to inflammation. These DAMPs are evolutionary conserved and have structural similarity to their bacterial ancestor. Therefore, cell-free mitochondria can act as a potent agent triggering the immune system in an autoimmune manner as well as a biomarker for cell damage and hypoxia.

Objective: The aim of this study is to investigate to role of epidural analgesia during birth, quantifying the copy number of circulating cell-free mitochondrial DNA in maternal serum and the placenta compared to controls. The investigators hypothesize that epidural analgesia with a local anesthetic has an effect on cell-free mitochondrial DNA levels, promoting the pathogenesis of ERMF and early inflammation. In addition, circulating mitochondrial DNA could be a potent biomarker for cell damage, early placenta hypoxia/insufficiency or preeclampsia.

Methods: For this study the investigators planned 3 groups each consisting of 15 patients. The intervention group (group 1) will be women with vaginal delivery having epidural analgesia and developing fever before delivery. The control group (group 2) will be women with vaginal delivery having an epidural analgesia without developing fever before delivery. Women with vaginal delivery without an epidural analgesia will serve as additional control (group 3). Blood will be taken at arrival at the delivery ward and immediately after delivery from a peripheral venous line. In addition, venous blood from the umbilical vein will be drawn postpartum. Axillary temperature will be measured routinely using a thermometer in a routine clinical fashion. Circulating cell-free mitochondrial DNA and other immunological markers will be quantified in maternal and umbilical cord (fetal) serum by real time quantitative PCR and statistical analysis will be performed by non-parametric tests.

ELIGIBILITY:
Inclusion Criteria:

* women
* between 18 and 45 years
* Para 0 or Para 1
* Gestational week
* Elective procedure 37±0 to 42±0

Exclusion Criteria:

* younger than 18 years
* Emergency procedures
* No written consent
* Fever <2 weeks
* Intraoperative conversion from one anesthetic or surgical procedure to another one.
* preeclampsia
* HELLP syndrome
* intrauterine growth reduction
* gestational diabetes mellitus
* autoimmune disease

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients must meet inclusion criteria and must give written consent. Informed consent will be obtained only for conscious patients preoperative. The cause of admission will be noted, baseline demographics and clinical history will be recorded. Patients included are giving birth at the Department of Obstetrics and Feto-Maternal Medicine at the Medical University of Vienna between July 2019 and July 2020. We are expecting to need to observe 15 patients per group in order to prove our hypothesis in this pilot study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
quantity of circulating cell-free mitochondrial DNA | change from quantity of baseline mtDNA to quantity of mtDNA immediately after delivery
  The aim of this study is to elucidate the influence of epidural analgesia (epidural analgesia or no epidural analgesia) during labor with regard to the quantity of circulating cell-free mitochondrial DNA in women developing ERMF.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesia, General Intensive Care and Pain Management,Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: Undecided